CLINICAL TRIAL: NCT04098172
Title: A Prospective, Multicenter Study to Evaluate the Performance and Safety of CometTM Pressure Guidewire in the Measurement of FFR in Chinese Patients
Brief Title: Evaluate the Performance and Safety of Comet Pressure Guidewire in the Measurement of FFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S2434
Record Dates: First submitted 2019-02-03; First posted 2019-09-23 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pressure Guidewire test subject (Experimental): Stable patients with suspected or known CAD, who are scheduled for diagnostic angiography and pressure wire assessment, and signed the informed consent, will be screened for enrollment in this study.
  Interventions: Device: Pressure Guidewire

INTERVENTIONS:
Device: Pressure Guidewire — Fractional Flow Reserve measurement

SUMMARY:
A prospective, open-label, multi-center study designed to validate the agreement of CometTM Pressure Guidewire and Pressure Wire Certus® in FFR measurements

DETAILED DESCRIPTION:
The COMET China study is a prospective, open-label, multi-center study designed to validate the agreement of CometTM Pressure Guidewire and Pressure Wire Certus® in FFR measurements. Patient with stable angina or any form of non-ST elevation acute coronary syndrome, who are scheduled for diagnostic angiography and pressure wire assessment, and signed the informed consent, will be screened for enrollment in this study.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient must be at least 18 years old and less than or equal to 75 years of age
2. Patient or his/her legally-authorized representative agrees to sign the EC-approved ICF prior to the procedure
3. Patient with stable angina or any form of non-ST elevation acute coronary syndrome and is clinically indicated of intra-coronary diagnostic angiography and FFR assessment

Angiographic Inclusion Criteria:

Moderate stenosis (30% to 70% diameter stenosis by visual estimation) is detected at diagnostic angiography

General Exclusion Criteria:

1. Patients unable to provide informed consent
2. Patients in pregnant state
3. Known renal insufficiency or failure (serum creatinine level of > 2.5 mg/dL, or on dialysis)
4. Allergy to the contrast
5. Significant arrhythmia, such as II degree or above of atrioventricular block, Sick sinus syndrome, ventricular tachycardia
6. Spastic bronchial asthma
7. ST elevation coronary syndrome
8. Hemodynamic instability
9. Contraindication to nitroglycerin or ATP
10. Current participation in another investigational drug or device clinical study that may affect the FFR measurements

Angiographic Exclusion Criteria:

CTO lesion Severe vessel tortuosity at the stenotic segments Culprit vessel of non-ST-segment elevation acute myocardial infarction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ning Guo, Dr, Principal Investigator — The First Afflilited Hospital of Xi,an Jiaotong University
Locations (2):
- China (2):
  - The First Affilited Hospital of Xi,an Jiaotong University, Xi'an, Shaanxi
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pressure Guidewire Test Subject
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pressure Guidewire Test Subject
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 8
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 58.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese han nationality | 39
Region of Enrollment [Number; unit: participants]
  China | 39
Weight [Geometric Mean (Standard Deviation); unit: Kg] | 70.9 (12.7)
Medical History [Count of Participants; unit: Participants]
  history of hypertension | 24
  history of diabetes | 9
  history of Cerebrovascular disease | 3
  history of Coronary heart disease | 37

OUTCOME MEASURES:

1. Primary Outcome: Fractional Flow Reserve (FFR)
Description: All eligible subjects will receive FFR measurements simultaneously by both CometTM Pressure Guidewire and Pressure wires Certus®. Fractional flow reserve (FFR) measurement involves determining the ratio between the maximum achievable blood flow in a diseased coronary artery and the theoretical maximum flow in a normal coronary artery. An FFR of 1.0 is widely accepted as normal. An FFR lower than 0.75-0.80 is generally considered to be associated with myocardial ischemia (MI).
  Agreement between the method of measurement will be confirmed if both conditions are met:
  The mean paired difference is within +/- 0.005
Time Frame: during procedure, 1 hour
Population: Pressure guide wire
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Comet Pressure Guidewire Test Subject; Certus Pressure Guidewire Test Subject: Stable patients with suspected or known Coronary Atherosclerotic Disease (CAD), who are scheduled for diagnostic angiography and pressure wire assessment, and signed the informed consent, will be screened for enrollment in this study.
  Pressure Guidewire: Fractional Flow Reserve measurement
Arm/Group | Comet Pressure Guidewire Test Subject | Certus Pressure Guidewire Test Subject
Number analyzed (Participants) | 39 | 39
Ratio | 0.862 [0.841 to 0.883] | 0.863 [0.842 to 0.884]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from subject procedure to subjects were discharged from hospital in 1 week.
Arm/Group | Pressure Guidewire Test Subject
All-Cause Mortality (participants affected / at risk) | 1/39
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pressure Guidewire Test Subject (N=39)
Subclavian artery stenosis (Vascular disorders) | 1 (39) — The SAE was not related to the study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT04098172/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT04098172/SAP_001.pdf